CLINICAL TRIAL: NCT05710666
Title: Single Arm Phase 2 Trial of Neoadjuvant Trastuzumab Deruxtecan (T-DXd) With Response-directed Definitive Therapy in Early Stage HER2-positive Breast Cancer: a Standard Chemotherapy-sparing Approach to Curative-intent Treatment - SHAMROCK Study
Brief Title: Neoadjuvant Trastuzumab Deruxtecan (T-DXd) With Response-directed Definitive Therapy in Early Stage HER2-positive Breast Cancer (SHAMROCK Study)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTRIAL-IE 22-01; 2022-002485-32 (EudraCT Number)
Record Dates: First submitted 2022-12-20; First posted 2023-02-02 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: HER2-positive Breast Cancer
MeSH Terms: interventions — trastuzumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- T-DXd (Experimental)
  Interventions: Drug: trastuzumab deruxtecan (T-DXd) (IV)

INTERVENTIONS:
Drug: trastuzumab deruxtecan (T-DXd) (IV) — Administered as an intravenous (IV) infusion at a dose of 5.4 mg/kg on Day 1 of each 21-day cycle for up to six cycles.

SUMMARY:
This study is a Phase 2 open label, single arm, adaptive multi-centre trial. Patients with early stage HER2-positive breast cancer will receive neoadjuvant treatment of trastuzumab deruxtecan (T-DXd) 5.4mg/kg intravenously every three weeks for up to six cycles.

DETAILED DESCRIPTION:
In this single arm Phase 2 trial we will administer T-DXd 5.4mg/kg intravenously every three weeks for up to six cycles. A mandatory repeat biopsy at Cycle 2 Day 14 +/- 4 days of starting T-DXd will be performed for the RNA Disruption Index (RDI) score assessment. As a safety measure patients will undergo clinical examination before each cycle of T-DXd to enable early identification of on-treatment locoregional progression. If progression is seen then T-DXd will be stopped and the patient will be taken off study treatment. In the absence of early progression, those patients with a high chance of pathological complete response (pCR) based on the RDI score will undergo repeat breast imaging after four cycles of T-DXd. Patients who have a high chance of pCR based on the RDI score will proceed to surgery after four cycles of T-DXd if they also have imaging complete response (iCR) at that point. Other patients who have a high chance of pCR based on the RDI score but iCR is not attained after four cycles or who have a low/intermediate chance of pCR based on the RDI score will undergo repeat breast imaging after six cycles of T-DXd. Patients with iCR after six cycles of T-DXd regardless of RDI score will proceed to surgery. Patients who have a low/intermediate chance of pCR based on the RDI score and residual disease on imaging after six cycles of T-DXd will undergo either further systemic therapy or proceed to surgery (at the discretion of their treating physician).

Based on the surgical specimen, patients who achieve a pCR will undergo further trastuzumab post-operatively to complete a total of 52 weeks of systemic therapy from the first cycle of T-DXd. Patients with residual disease at surgery will receive adjuvant chemotherapy as decided by the treating physician.

ELIGIBILITY:
Inclusion Criteria:

1. Adult women and men ≥ 18 years of age.
2. Histologically confirmed HER2-positive breast cancer:

   o Documented HER2 overexpression by local laboratory (IHC 3+ or FISH or CISH positive on diagnostic breast biopsy).
3. Newly diagnosed breast cancer, planned for neoadjuvant therapy prior to surgery.
4. Stages 2-3 breast cancer.
5. Patients should not have received any prior therapy for breast cancer.
6. Patients must be willing to undergo mandatory tumour biopsy at Cycle 2 Day 14 (+/- 4 days) and (if applicable, refer to section 9.5 Tomosynthesis-Guided Core Biopsies sub-study and Table 8-2) before surgery .
7. ECOG performance status 0-1.
8. Availability of archival tumour biopsy tissue at screening.
9. Left ventricular ejection fraction (LVEF) ≥ 50%, as determined by ECHO or MUGA.
10. Adequate laboratory values collected no more than 14 days before registration. All parameters must meet the inclusion criteria on the same day, and must be the most recent results available:

    * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L (granulocyte-colony stimulating factor administration is not allowed within 1 week prior to C1D1)
    * Platelet count ≥ 100 x 109/L (Platelet transfusion is not allowed within 1 week prior to C1D1)
    * Haemoglobin ≥ 9.0 g/dL. NOTE: Participants requiring ongoing transfusions or growth factor support to maintain haemoglobin ≥9.0 g/dL are not eligible (Red blood cell transfusion is not allowed within 1 week prior to C1D1).
    * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 × upper limit of normal (ULN)
    * Total bilirubin ≤ 1.5xULN or < 3×ULN in the presence of documented Gilbert's syndrome (unconjugated hyperbilirubinemia)
    * Serum albumin ≥ 25 g/L
    * Creatinine clearance (CrCL) ≥ 30ml/min as determined by Cockcroft Gault (using actual body weight) (refer to Appendix C).
    * Prothrombin time and either partial thromboplastin or activated partial thromboplastin time ≤ 1.5 × ULN.
11. Evidence of post-menopausal status or negative serum pregnancy test for females of childbearing potential who are sexually active with a non-sterilized male partner. For women of childbearing potential, a negative result for serum pregnancy test must be available at the screening visit.

    Women of childbearing potential are defined as those who are not surgically sterile (i.e. underwent bilateral salpingectomy, bilateral oophorectomy, or complete hysterectomy) or post-menopausal. Postmenopausal women defined as:

    i. Women aged <50 years will be considered post-menopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels in the post-menopausal range for the site.

    ii. Women aged ≥50 years will be considered post-menopausal if they have been amenorrhoeic for 12 months or more following cessation of all exogenous hormonal treatments.

    iii. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods outlined for women of child-bearing potential if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to registration. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.
12. Women of childbearing potential must agree to use a highly effective method of contraception according to current HMA CTFG guideline when sexually active. This applies from signing of the informed consent form until at least 7 months after the last IMP administration. The investigator or a designated associate is required to advise the patient how to achieve an adequate birth control. Highly effective contraception is defined in the study as methods that achieve a failure rate of less than 1% per year when used consistently and correctly. Such methods include:

    i. Combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal).

    ii. Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable and implantable).

    iii. Intrauterine device (IUD). iv. Intrauterine hormone-releasing system (IUS). v. Bilateral tubal occlusion. vi. Successfully vasectomised partner. vii. Sexual abstinence.
13. Non-sterilized male patients who are sexually active with a female partner of childbearing potential must use a condom with spermicide from screening to 4 months after the final dose of IMP. Complete heterosexual abstinence for the duration of the study and drug washout period is an acceptable contraceptive method if it is in line with the patient's usual lifestyle (consideration must be made to the duration of the clinical trial); however, periodic or occasional abstinence, the rhythm method, and the withdrawal method are not acceptable. It is strongly recommended for the female partners of a male patient to also use at least one highly effective method of contraception throughout this period. In addition, male patients should refrain from fathering a child, or freezing or donating sperm from the time of registration, throughout the study and for 4 months after the last dose of IMP. Preservation of sperm should be considered prior to enrollment in this study.
14. Female patients must not donate, or retrieve for their own use, ova from the time of registration and throughout the study treatment period, and for at least 7 months after the final IMP administration. They should refrain from breastfeeding throughout this time. Preservation of ova may be considered prior to enrollment in this study.

Exclusion Criteria:

1. Known metastatic or stage 4 breast cancer.
2. Unstable angina (angina symptoms at rest), new-onset angina (begun within the last 3 months). Myocardial infarction (MI) less than 6 months before registration, symptomatic congestive heart failure (CHF) (New York Heart Association Class II to IV). Patients with troponin levels above ULN at screening and without any myocardial related symptoms, should have a cardiologic consultation before enrollment to rule out MI.
3. Corrected QT interval (QTcF) prolongation to >470 msec (females) or >450 msec (males) based on the screening 12-lead ECG.
4. Uncontrolled arterial hypertension despite optimal medical management (per investigator's opinion).
5. Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 3 months before registration.
6. Non-healing wound, ulcer, or bone fracture.
7. Active, clinically serious infections > CTCAE Grade 2 (CTCAE v5.0) requiring IV antibiotics, antivirals, or antifungals.
8. Patients with evidence or history of bleeding diathesis. Any haemorrhage or bleeding event ≥ CTCAE Grade 3 within 4 weeks prior to the start of study treatment.
9. Active primary immunodeficiency, known human immunodeficiency virus (HIV) infection, or active hepatitis B or C infection. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
10. History of (non-infectious) ILD/pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening.
11. Lung criteria:

    1. Lung-specific intercurrent clinically significant illnesses including, but not limited to, any underlying pulmonary disorder (e.g. pulmonary emboli within three months before study registration, severe asthma, severe COPD, restrictive lung disease, pleural effusion, etc.)
    2. Any autoimmune, connective tissue or inflammatory disorders (e.g. Rheumatoid arthritis, Sjogren's, sarcoidosis etc.) where there is documented, or a suspicion of pulmonary involvement at the time of screening. Full details of the disorder should be recorded in the eCRF for patients who are included in the study.
    3. Prior pneumonectomy (complete)
12. Receipt of live, attenuated vaccine (mRNA and replication deficient adenoviral vaccines are not considered attenuated live vaccines) within 30 days prior to the first dose of trastuzumab deruxtecan. Note: Patients, if enrolled, should not receive live vaccine during the study and up to 30 days after the last dose of IMP.
13. Pregnant or breast-feeding female patients, or patients who are planning to become pregnant.
14. Concomitant use of prohibited medications (refer to section 7.6.3: Prohibited Concomitant Medications and Treatments).
15. Known hypersensitivity to the test drug, test drug class, or excipients in the formulation.
16. History of severe hypersensitivity reactions to other monoclonal antibodies.
17. Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.
18. Any illness or medical conditions that are unstable or could jeopardize the safety of patients and their compliance in the study.
19. Multiple primary malignancies within 3 years before study registration, with the exception of

    1. adequately resected non-melanoma skin cancer
    2. curatively treated in-situ disease
    3. other solid tumours curatively treated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2023-10-26 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients who achieve pCR after T-DXd treatment | From registration until surgery, approximately 18 weeks
  The percentage of patients who achieve pCR after T-DXd treatment and thus avoid standard cytotoxic chemotherapy

SECONDARY OUTCOMES:
pCR rate in all other patients (patients who could not avoid standard cytotoxic chemotherapy) and in the entire study population. | From registration until surgery, approximately 18 weeks
3-year EFS of patients treated with only T-DXd and trastuzumab. | 3 years from registration
  EFS is defined as time from registration to disease recurrence, progression or death from any cause.
3-year overall survival (OS) of patients treated with only T-DXd and trastuzumab. | 3 years from registration
  OS is defined as the time from registration to date of death from any cause, censored at date last known to be alive for those who have not died.
3-year EFS of patients treated with systemic therapy other than trastuzumab in addition to T-DXd. | 3 years from registration
3-year OS of patients treated with systemic therapy other than trastuzumab in addition to T-DXd. | 3 years from registration
3-year EFS and OS of the entire study population. | 3 years from registration
3-year OS of the entire study population. | 3 years from registration
3-year EFS difference between patients achieving vs not achieving pCR at surgery. | 3 years from registration
3-year OS difference between patients achieving vs not achieving pCR at surgery. | 3 years from registration
Molecular evolution of tumours during treatment assessed by ctDNA. | From registration until end of study treatment, approximately 23 weeks
Molecular evolution of tumours during treatment assessed by protein biomarkers. | From registration until end of study treatment, approximately 23 weeks
Molecular evolution of tumours during treatment assessed by CTCs analysis. | From registration until end of study treatment, approximately 23 weeks
Percentage of patients who achieve pCR after 4 cycles of T-DXd. | From registration until surgery, approximately 18 weeks
The sensitivity and specificity for prediction of pCR of RDI and imaging and tomosynthesis biopsy alone and in combination. | From registration until surgery, approximately 18 weeks

CONTACTS AND LOCATIONS:
Locations (5):
- Ireland (5):
  - University Hospital Galway, Galway, Connacht
  - Saint Vincent's University Hospital, Dublin, Leinster
  - Beaumont Hospital, Dublin, Leinster
  - Cork University Hospital, Cork, Munster
  - University Hospital Limerick, Limerick, Munster

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dowling GP, Toomey S, Bredin P, Parker I, Mulroe E, Marron J, McLoughlin O, Teiserskiene A, Power C, O'Shea AM, Greally M, Morris PG, Duke D, Hill ADK, Hennessy BT. Neoadjuvant trastuzumab deruxtecan (T-DXd) with response-directed definitive therapy in early stage HER2-positive breast cancer: a phase II study protocol (SHAMROCK study). BMC Cancer. 2024 Jan 17;24(1):91. doi: 10.1186/s12885-024-11851-4. PMID 38233810